CLINICAL TRIAL: NCT05426031
Title: Optimal Protamine Dosing for Heparin Reversal Following Cardiopulmonary Bypass: A Blinded Randomized Control Trial Comparing Two Strategies
Brief Title: Optimal Protamine Dosing for Heparin Reversal Following Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michael Fabbro, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220234
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Coagulation; Intravascular
MeSH Terms: conditions — Thrombosis | interventions — Protamines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed Dose Protamine group (Experimental): Participants in the group will receive a one time dose of 250 mg Protamine to reverse heparin during the standard cardiopulmonary bypass management during cardiac surgery.
  Interventions: Drug: Protamine fixed dose
- Ratio Dose Protamine Group (Active Comparator): Participants in the group will receive a ratio dose of Protamine in a 1mg per 100 units of heparin ratio to reverse heparin during the standard cardiopulmonary bypass management during cardiac surgery.
  Interventions: Drug: Protamine ratio dose

INTERVENTIONS:
Drug: Protamine fixed dose — 250 mg of protamine intravenously (IV), one time use
  Arms: Fixed Dose Protamine group
Drug: Protamine ratio dose — 1mg of protamine per 100 units of heparin given intravenously (IV), one time use
  Arms: Ratio Dose Protamine Group

SUMMARY:
The purpose of this study is to compare two different dosing strategies of a drug named protamine.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age undergoing elective cardiac surgery with cardiopulmonary bypass.
* Patients must that have a calculated protamine dose greater than 250 mg based on standard 1:1 initial heparin to protamine dosing calculation.

Exclusion Criteria:

* Patients who are under 18 years of age or pregnant.
* Patients undergoing emergency surgery (ASA class E).
* Patients with known coagulation disorders.
* Patients requiring circulatory arrest or deep hypothermia.
* Patients who have not had the appropriate interruption in coumadin, direct oral anticoagulants or non-aspirin antiplatelet agents.
* Patients on pre-operative intravenous unfractionated heparin infusions.
* Patients ineligible for heparin administration due to known adverse reactions including allergy or heparin induced thrombocytopenia or known heparin resistance.
* Patients who are unable to provide informed consent in the form of a signature.
* History of adverse reaction to protamine.
* Have any condition that, in the opinion of the investigator, will compromise the well-being of the patient or the study, or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fabbro, DO, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Hospital, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Started | 65 | 65
Completed | 62 | 63
Not Completed | 3 | 2
Not completed — Circulatory Arrest | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 40 | 66
  >=65 years | 39 | 25 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.5 [58 to 74] | 63 [53 to 70] | 64.7 [53 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 51 | 51 | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Activated Clotting Time
Description: Activated clotting times will be measured using standard coagulation monitor
Time Frame: Baseline (before start of surgery)
Population: Data was collected for all subjects that completed
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Number analyzed (Participants) | 62 | 63
seconds | 116 [108 to 122] | 113 [107 to 121]

2. Primary Outcome: Activated Clotting Time
Description: Activated clotting times will be measured using standard coagulation monitor
Time Frame: up to 4 hours (after cardiopulmonary bypass surgery)
Population: Data was collected for all subjects that completed
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Number analyzed (Participants) | 62 | 63
seconds | 121.5 [114 to 133] | 120.5 [114 to 135]

3. Secondary Outcome: Additional Protamine Dosing
Description: Additional protamine dose will be measured in milligrams (mg)
Time Frame: Up to 4 hours
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Number analyzed (Participants) | 62 | 63
milligrams | 0 [0 to 30] | 0 [0 to 25]

4. Secondary Outcome: Chest Tube Output
Description: Measured in milliliters (ml)
Time Frame: Up to 24 hours
Population: Data was collected for all subjects that completed
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Number analyzed (Participants) | 62 | 63
ml | 640 [500 to 760] | 640 [535 to 840]

5. Secondary Outcome: Count of Participants Receiving Red Blood Cell Transfusion
Description: All transfusions were recorded in a data log for the count of participants that received a red blood cell transfusion.
Time Frame: Up to 4 hours
Population: Data was collected for all subjects that completed
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
Number analyzed (Participants) | 62 | 63
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Fixed Dose Protamine Group | Ratio Dose Protamine Group
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05426031/Prot_SAP_000.pdf